CLINICAL TRIAL: NCT00570908
Title: A Phase 2 Trial of Capecitabine Concomitantly With Whole Brain Radiotherapy(WBRT) Followed by Capecitabine and Sunitinib for Central Nervous System, (CNS) Metastases in Breast Cancer
Brief Title: Brain Mets - Capecitabine Plus Sunitinib and WBRT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to poor accrual this study is being closed to accrual
Sponsor: Baylor Breast Care Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-20924; H 20924 (Other: Baylor College of Medicine)
Record Dates: First submitted 2007-12-07; First posted 2007-12-11 (Estimated); Results first posted 2014-08-12 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-08

CONDITIONS: Breast Cancer
Keywords: brain metastasis; breast cancer; metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms; Brain Neoplasms | interventions — Sunitinib; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Study Group (Experimental): capecitabine administered concurrently with WBRT followed by combination the combination of capecitabine with sunitinib
  Interventions: Drug: sunitinib; Drug: capecitabine; Radiation: WBRT

INTERVENTIONS:
Drug: sunitinib — Sutent
Drug: capecitabine — concurrently
Radiation: WBRT — Whole Brain Radiotherapy 30 Gy in 10 fractions
  Other Names: Whole Brain Radiotherapy

SUMMARY:
The purpose of this study is to assess the efficacy and safety of concurrent whole brain radiotherapy (WBRT) and capecitabine followed by combination capecitabine and sunitinib in treating patients with CNS metastases from breast cancer.

DETAILED DESCRIPTION:
Central nervous system (CNS) metastases is the most common type of brain malignancy, and breast cancer is the second most common type of malignancy to cause CNS metastases. Although the incidence of CNS metastases is less common than bone or visceral metastases, it is associated with poorer prognosis and is relatively unresponsive to systemic therapies. The incidence of CNS metastases in breast cancer has been estimated as 1-16% in clinical series, with higher rates (18-30%) in autopsy series. Recently a trend towards increasing CNS relapse has been noted, up to 25-34%. This may be partly explained by the increasing use of contrast-enhanced magnetic resonance imaging (MRI), heightened awareness by patient or clinicians, or an alteration in the natural history of breast cancer with improvements in systemic therapies, resulting in a prolongation of survival. Therefore, with improvements in treatments, metastases are better controlled, resulting in the CNS becoming a sanctuary for residual disease. The treatment of CNS metastases in breast cancer remains challenging. Surgical resection of tumor will prolong survival only in patients with a single lesion and with well controlled systemic disease. For patients with multiple lesions, whole brain radiotherapy (WBRT) remains the backbone in the management of CNS metastases. Recently the use of stereotactic radiosurgery alone or in combination with WBRT has been explored. Although better local control was achieved with the combination therapy, minimal overall survival benefit was seen. This may be secondary to the competing risk of death from systemic (extra-CNS) progression. The use of systemic agents including chemotherapy and hormonal therapy has been generally disappointing. This is often attributed to the impermeability of the blood-brain and blood-tumor barriers. Furthermore, P-glycoprotein (Pgp), a drug efflux pump encoded by the multidrug resistance gene, mdR1, is expressed in brain endothelial cells. Therefore, agents such as doxorubicin, cyclophosphamide, 5-fluorouracil, paclitaxel, docetaxel and vinorelbine, which are active against breast cancer, may either penetrate CNS poorly, or be transported out of the CNS environment. However, the blood brain barrier may be more leaky and permeable than previously thought in patients with CNS metastases, and these agents may achieve therapeutic concentrations in the CNS. As evidence for this, patients without prior exposure to agents such as cyclophosphamide, methotrexate, 5-fluorouracil, vincristine, and doxorubicin, can have significant objective responses in the CNS metastases. Today, most patients would have received these agents in the adjuvant setting, thus emphasizing the importance of both chemo-sensitivity together with CNS penetration, in the treatment of CNS metastases.

This is a single arm, open label, phase II drug study. This study will be conducted at the Breast Care Center at Baylor College of Medicine and its affiliated hospital, and at Ben Taub General Hospital in Houston. Patients who were diagnosed with CNS metastases (brain +/- leptomeningeal disease) will be identified prospectively. All eligible patients will receive capecitabine concurrently with WBRT followed by combination capecitabine with sunitinib. WBRT will be administered at 30 Gy in 10 fractions together with capecitabine to be given on the first day of WBRT at 1000 mg/m2/day and continued daily for 14 days. After a 7 days rest period, capecitabine will be restarted at 2000mg/m2/day for 14 days followed by a 7 days rest period. This will be given together with sunitinib at 37.5 mg daily. This is the dosing determined by the phase I study with capecitabine and sunitinib. Dose reduction and/or treatment postponement will be done for significant toxicity. Capecitabine with sunitinib will be administered until disease progression in either CNS and/or non-CNS sites. Efficacy assessments will be performed on all subjects via imaging studies in the CNS and extra-CNS sites 8 weeks after starting study, then every 12 weekly. Neurological examination will be performed at baseline, 3 weeks after starting treatment, then every 6 weekly. Assessment of treatment toxicity will be performed at baseline, 3 weeks after starting treatment, then every 3 weekly using the NCI Common Toxicity grading system. Clinical and laboratory parameters will be assessed until disease progression or withdrawal from study (due to unacceptable toxicity or withdrawal of consent). Subjects with progression of CNS and / or extra-CNS disease will be considered progressors. Subjects withdrawn from treatment will be followed for survival until death.

Primary endpoint: 1. To determine progression free survival. Progression will be defined by progression in either CNS or extra-CNS metastases. Secondary endpoint: 1. To assess the toxicities associated with the regimen 2. To determine the overall objective response in CNS disease 3. To determine the overall objective response in extra-CNS disease 4. To determine the overall survival.

ELIGIBILITY:
Inclusion Criteria:

Patients must be age 18 or older. Histological or cytologically confirmed invasive breast cancer, with Stage IV disease.

Evidence of radiographically measurable CNS metastases (greater than or equal to 10mm on T1-weighted gadolinium-enhanced MRI) within 2 weeks prior to starting treatment. Patients without known extra-CNS disease are eligible.

Must have metastases in the brain. Patients with concurrent leptomeningeal carcinomatosis are eligible for the study. Local radiation to sites of meningeal involvement in the spine is allowed.

No prior whole brain radiation. Patients who had previous stereotactic brain irradiation are eligible, provided they have new measurable brain lesions (which has not been radiated previously) and will receive WBRT at 30Gy over 10 fractions.

May undergo surgical resection of CNS metastases if clinically indicated, but must have remaining measurable disease in the brain after surgery.

No prior treatment with capecitabine in the adjuvant or metastatic settings. Patients may have completed 5-fluorouracil based treatment in the adjuvant setting or metastatic setting more than one year prior.

Patients who had previous trastuzumab therapy will be eligible but treatment will be discontinued prior to enrollment.

Cardiac ejection fraction within institutional range of normal as measure by echocardiogram or MUGA scans at baseline.

Hematological adequacy Hepatic adequacy Renal adequacy Must have recovered from toxicity of prior chemotherapy with laboratory values as specified above. Concurrent treatment with bisphosphonates is permitted. Performance status of ECOG 0-1.

Life expectancy of at least 12 weeks. At least 3 weeks since major surgical procedures. Able to swallow and retain oral medication.

Exclusion Criteria:

Pregnant or breast feeding. Known allergy to capecitabine or 5-fluorouracil. Known to have dihydropyrimidine dehydrogenase (DPD) deficiency.

Patients who have leptomeningeal carcinomatosis as the only site of CNS metastases.

Patients taking concomitant medications which are CYP3A4 inhibitors or inducers.

Patients who will receive intrathecal chemotherapy for leptomeningeal disease. Patients with psychiatric or addictive disorders that would adversely effect compliance with oral medication.

Life expectancy less than 3 months. Symptomatic lymphangitic spread to lung. Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel.

History of immediate or delayed hypersensitivity reaction to gadolinium contrast agents, or other contraindication or gadolinium contrast.

Other known contraindication to MRI, such as a cardiac pacemaker, implanted cardiac defibrillator, brain aneurysm clips, cochlear implant, ocular foreign body, or shrapnel,

1Vascular disease within 12 months prior to enrollment Uncontrolled infection History of other malignancy, except for curatively treated basal cell carcinoma or squamous cell carcinoma of the skin, or carcinoma in situ of the cervix. Subjects with other malignancies who have been disease-free for at least 5 years are eligible

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-02; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mothaffar' Rimawi, MD, Principal Investigator — Baylor College of Medicine, Breast Center
Locations (1):
- Lester and Sue Smith Breast Center at Baylor College of Medicine, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- WBRT + Capecitabine + Sunitinib: capecitabine concurrently with WBRT(Whole Brain Radiotherapy 30 Gy in 10 fractions) followed by combination capecitabine with sunitinib(Sutent)
Period: Overall Study
Arm/Group | WBRT + Capecitabine + Sunitinib
Started | 12
Completed | 5 (5 patients progressed during the study treatment)
Not Completed | 7
Not completed — Adverse Event | 5
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: 12 patients were enrolled and started treatment
Arm/Group | WBRT + Capecitabine + Sunitinib
Number analyzed (Participants) | 12
Age, Continuous [Median (Full Range); unit: years] | 50 [32 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Progression free survival is defined as form initiation of WBRT with capecitabine to the time of first documented progression at any site (CNS or non-CNS site) or death due to any cause, where progression is defined stringently by progression in either CNS or extra-CNS metastases.
Time Frame: 2 years
Population: 5 patients progressed during the study treatment. 7 patients were off study treatment early due to AE or withdrawal but 6 of them were followed for the survival outcome, 1 was lost to follow up after 3.5 months observation (censored data).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | WBRT + Capecitabine + Sunitinib
Number analyzed (Participants) | 12
months | 4.7 [2.1 to 7.1]

ADVERSE EVENTS:
Arm/Group | WBRT + Capecitabine + Sunitinib
Serious Adverse Events (participants affected / at risk) | 4/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | WBRT + Capecitabine + Sunitinib (N=12)
Cardiac - CHF (Cardiac disorders) | 1 (1)
Dyspnea (SOB) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Diabetetic Ketoacidosis (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | WBRT + Capecitabine + Sunitinib (N=12)
Alkaline Phosphate (Metabolism and nutrition disorders) | 3 (4)
AST (Metabolism and nutrition disorders) | 6 (11)
Bilirubin, Elevated (Metabolism and nutrition disorders) | 3 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dehydration (Gastrointestinal disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Fatifue (General disorders) | 8 (10)
Hand-Foot Skin Reaction (Skin and subcutaneous tissue disorders) | 5 (7)
Hemoglobin (Blood and lymphatic system disorders) | 4 (7)
Hyperbilirubinemia (Metabolism and nutrition disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 5 (6)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2)
Leukocytes (Metabolism and nutrition disorders) | 5 (7)
Mood Alteration - Depression (Psychiatric disorders) | 3 (3)
Mucositis - Oral (Gastrointestinal disorders) | 6 (8)
Nausea (Gastrointestinal disorders) | 7 (8)
Neutropenia (Infections and infestations) | 2 (2)
Pain - Headache (Nervous system disorders) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 (10)
TSH (Endocrine disorders) | 2 (2)
vomiting (Gastrointestinal disorders) | 2 (2)
ALT (Metabolism and nutrition disorders) | 1 (1)
ANC low (Blood and lymphatic system disorders) | 1 (1)
Anorexia (Gastrointestinal disorders) | 1 (1)
Bilateral Pedal Edema (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dry Mouth (Gastrointestinal disorders) | 1 (1)
Dysgeusia (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Erythema - Right Axillary (Skin and subcutaneous tissue disorders) | 1 (1)
E. Coli Bacteremia (Infections and infestations) | 1 (1)
Fever (General disorders) | 1 (1)
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Gums - Bleeding (Blood and lymphatic system disorders) | 1 (1)
Hemolysis (Blood and lymphatic system disorders) | 1 (1)
Hypernaturia (Metabolism and nutrition disorders) | 1 (1)
Infection - Middle Ear (Infections and infestations) | 1 (1)
Infection - Sinus (Infections and infestations) | 1 (1)
Oral Thrush (Gastrointestinal disorders) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (2)
Rash - Leg (Skin and subcutaneous tissue disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1)
Urinary Frequency (Renal and urinary disorders) | 1 (1)
Vision - Flashing Lights (Eye disorders) | 1 (1)
Low WBC (Blood and lymphatic system disorders) | 1 (1)
Yellow skin (Skin and subcutaneous tissue disorders) | 1 (1)
Pain (General disorders) | 6 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes